CLINICAL TRIAL: NCT05803018
Title: A Phase Ib/II Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Efficacy of BL-B01D1 for Injection in Patients With Multiple Solid Tumors, Including Recurrent or Metastatic Gynecological Malignancies
Brief Title: A Study of BL-B01D1 in Patients With Multiple Solid Tumors, Including Recurrent or Metastatic Gynecological Malignancies
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sichuan Baili Pharmaceutical Co., Ltd. (Industry)
Collaborators: Baili-Bio (Chengdu) Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BL-B01D1-202
Record Dates: First submitted 2023-03-23; First posted 2023-04-07 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Gynecological Malignant Tumor; Solid Tumor
Keywords: Ovarian Cancer; Endometrial Carcinoma; Cervical Cancer; Tubal carcinoma
MeSH Terms: conditions — Ovarian Neoplasms; Endometrial Neoplasms; Uterine Cervical Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study treatment (Experimental): Participants receive BL-B01D1 as intravenous infusion for the first cycle (3 weeks). Participants with clinical benefit could receive additional treatment for more cycles. The administration will be terminated because of disease progression or intolerable toxicity occurring or other reasons.
  Interventions: Drug: BL-B01D1

INTERVENTIONS:
Drug: BL-B01D1 — Administration by intravenous infusion
  Other Names: iza-bren; izalontamab brengitecan; BMS-986507

SUMMARY:
A phase Ib/II clinical study to evaluate the safety, tolerability, pharmacokinetics and efficacy of BL-B01D1 for injection in patients with multiple solid tumors, including recurrent or metastatic gynecological malignancies.

DETAILED DESCRIPTION:
Phase Ib: To explore the safety and initial efficacy of BL-B01D1 in a variety of solid tumors, including recurrent or metastatic gynecological malignancies, to further identify RP2D. To evaluate the initial efficacy of BL-B01D1. The pharmacokinetic characteristics and immunogenicity of BL-B01D1 were further evaluated. Phase II: To explore the efficacy of BL-B01D1 as a single agent RP2D in patients with multiple solid tumors such as recurrent or metastatic gynecological malignancies using Phase Ib clinical studies. To evaluate the safety and tolerance of BL-B01D1. To evaluate the pharmacokinetic characteristics and immunogenicity of BL-B01D1.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily sign the informed consent form and comply with the protocol requirements;
2. Age: ≥18 years and ≤75 years;
3. Expected survival time ≥3 months;
4. Histologically and/or cytologically confirmed recurrent or metastatic gynecological malignancies with failed standard treatment, intolerance to standard treatment, or no current standard treatment available;
5. Agree to provide archived tumor tissue specimens (10 slides) or fresh tissue samples from primary or metastatic lesions within the past 3 years;
6. Must have at least one measurable lesion as defined by RECIST v1.1;
7. ECOG performance status score of 0 or 1;
8. Toxicity from prior anti-tumor therapy has recovered to ≤ Grade 1 as defined by NCI-CTCAE v5.0;
9. No severe cardiac dysfunction, with left ventricular ejection fraction (LVEF) ≥50%;
10. Organ function levels must meet the requirements without transfusion, albumin, colony-stimulating factors, any cell growth factors, and/or platelet-raising drugs within 14 days before the first dose of the study drug;
11. Coagulation function: International Normalized Ratio (INR) ≤1.5, and activated partial thromboplastin time (APTT) ≤1.5 × ULN;
12. Urine protein ≤2+ or ≤1000 mg/24h;
13. For premenopausal women with childbearing potential, a pregnancy test (serum or urine) must be performed within 7 days before starting treatment, and the result must be negative; they must not be breastfeeding. All enrolled patients must use adequate barrier contraception throughout the treatment period and for 6 months after treatment ends.

Exclusion Criteria:

1. Received chemotherapy, biological therapy, immunotherapy, or other antitumor treatments within 4 weeks or 5 half-lives prior to the first dose (6 weeks for mitomycin and nitrosoureas; oral fluorouracil drugs, etc.);
2. History of severe heart disease;
3. Prolonged QT interval, complete left bundle branch block, third-degree atrioventricular block, or severe arrhythmia;
4. Active autoimmune or inflammatory diseases;
5. Other malignancies with progression or requiring treatment within 5 years prior to the first dose;
6. Poorly controlled hypertension (systolic blood pressure >150 mmHg or diastolic blood pressure >100 mmHg) despite the use of two antihypertensive medications;
7. Poorly controlled blood glucose levels;
8. History of interstitial lung disease (ILD), current ILD, or suspected ILD based on imaging during screening;
9. Concurrent pulmonary disease leading to clinically significant respiratory impairment;
10. Unstable thrombotic events requiring therapeutic intervention within 6 months before screening;
11. Patients with central nervous system (CNS) metastases and/or carcinomatous meningitis (leptomeningeal metastases);
12. Patients with significant serous cavity effusion, symptomatic effusion, or poorly controlled effusion;
13. History of hypersensitivity to recombinant humanized antibodies or human-mouse chimeric antibodies, or any excipients of BL-B01D1;
14. Imaging findings indicating tumor invasion or encasement of major thoracic, cervical, or pharyngeal blood vessels;
15. Previous organ transplantation or allogeneic hematopoietic stem cell transplantation (Allo-HSCT);
16. Cumulative anthracycline dose >360 mg/m² in prior (neo)adjuvant anthracycline therapy;
17. Positive for human immunodeficiency virus (HIV) antibodies, active tuberculosis, active hepatitis B virus (HBV) infection, or active hepatitis C virus (HCV) infection;
18. Severe infection within 4 weeks before the first dose of the study drug; signs of active pulmonary infection within 2 weeks before the first dose;
19. Participation in another clinical trial within 4 weeks before the first dose;
20. Any other condition deemed unsuitable for participation in this clinical trial by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2023-06-25 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Phase Ib: Recommended Phase II Dose (RP2D) | Up to approximately 24 months
  The RP2D is defined as the dose level chosen by the sponsor (in consultation with the investigators) for phase II study, based on safety, tolerability, efficacy, PK, and PD data collected during the dose escalation study of BL-B01D1.
Phase II: Objective response rate (ORR) | Up to approximately 24 months
  ORR is defined as the percentage of participants, who has a CR (disappearance of all target lesions) or PR (at least a 30% decrease in the sum of diameters of target lesions). The percentage of participants who experiences a confirmed CR or PR is according to RECIST 1.1.

SECONDARY OUTCOMES:
Phase Ib/II: Treatment-Emergent Adverse Event (TEAE) | Up to approximately 24 months
  TEAE is defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally emerging, or any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a pre-existing condition during the treatment of BL-B01D1. The type, frequency and severity of TEAE will be evaluated during the treatment of BL-B01D1.
Phase Ib: Objective response rate (ORR) | Up to approximately 24 months
  ORR is defined as the percentage of participants, who has a CR (disappearance of all target lesions) or PR (at least a 30% decrease in the sum of diameters of target lesions). The percentage of participants who experiences a confirmed CR or PR is according to RECIST 1.1.
Phase II: Progression-free survival (PFS) | Up to approximately 24 months
  The PFS is defined as the time from the participant's first dose of BL-B01D1 to the first date of either disease progression or death, whichever occurs first.
Phase Ib/II: Disease control rate (DCR) | Up to approximately 24 months
  The DCR is defined as the percentage of participants who has a CR, PR, or Stable Disease (SD: neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease [PD: at least a 20% increase in the sum of diameters of target lesions and an absolute increase of at least 5 mm. The appearance of one or more new lesions is also considered PD]).
Phase Ib/II: Duration of response (DOR) | Up to approximately 24 months
  The DOR for a responder is defined as the time from the participant's initial objective response to the first date of either disease progression or death, whichever occurs first.
Phase Ib/II: Cmax | Up to approximately 24 months
  Maximum serum concentration (Cmax) of BL-B01D1 will be investigated.
Phase Ib/II: Tmax | Up to approximately 24 months
  Time to maximum serum concentration (Tmax) of BL-B01D1 will be investigated.
Phase Ib: T1/2 | Up to approximately 24 months
  Half-life (T1/2) of BL-B01D1 will be investigated.
Phase Ib: AUC0-t | Up to approximately 24 months
  Blood concentration - Area under time line.
Phase Ib: CL | Up to approximately 24 months
  To study the serum clearance rate of BL-B01D1 per unit time.
Phase Ib/II: Ctrough | Up to approximately 24 months
  Ctrough is defined as the lowest serum concentration of BL-B01D1 prior to the next dose will be administered.
Phase Ib/II: Anti-drug antibody (ADA) | Up to approximately 24 months
  Frequency and titer of anti-BL-B01D1 antibody (ADA) will be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaohua Wu, PHD, Principal Investigator — Fudan University; Jian Zhang, PHD, Principal Investigator — Fudan University
Locations (1):
- Fudan University ShangHai Cancer Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No